CLINICAL TRIAL: NCT05857748
Title: Examining the Clinical Characteristics, Treatment Patterns, Real-world Effectiveness, and Healthcare Resource Utilization of Patients With Dry Eye Disease Receiving Lifitegrast Ophthalmic Solution in the United Arab Emirates: a Prospective Cohort
Brief Title: Examining the Clinical Characteristics, Treatment Patterns, Real-world Effectiveness, and Healthcare Resource Utilization of Patients With Dry Eye Disease
Status: Withdrawn | Type: Observational
Why Stopped: Company decision due to the transfer of ownership of the product
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLIF606A1AE01
Record Dates: First submitted 2023-04-27; First posted 2023-05-15 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Dry Eye Disease
Keywords: Dry eye disease; DED; NIS; United Arab Emirates
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Single arm of DED patients: 1. Age ≥18 years at index date.
  2. Confirmed diagnosis of DED.
  3. Newly started on lifitegrast ophthalmic solution within the recruitment period and not receiving lifitegrast ophthalmic solution within 6 months prior to recruitment.
  4. Received continuous medical care at the healthcare site defined as at least one clinical visit within 6 months.
  Interventions: Drug: lifitegrast

INTERVENTIONS:
Drug: lifitegrast — patient newly started on medication will be followed for 6 months

SUMMARY:
A prospective, non- interventional, observational, non-comparative, longitudinal cohort study design will be used to address the objectives of this study using data collected through a healthcare.

DETAILED DESCRIPTION:
The study will identify patients with DED who newly initiated treatment with lifitegrast ophthalmic solution on or after the start of the recruitment period, which will last for 1 year since first patient first visit (FPFV) (index period). A minimum follow-up period of 6 months (post-index period) is set for each patient making the last patient last visit (LPLV) 6 months after the closure of recruitment period or after the last patient recruited, whichever comes first.

ELIGIBILITY:
Inclusion criteria

1. Age ≥18 years at index date.
2. Confirmed diagnosis of DED.
3. Newly started on lifitegrast ophthalmic solution within the recruitment period and not receiving lifitegrast ophthalmic solution within 6 months prior to recruitment.
4. Received continuous medical care at the healthcare site defined as at least one clinical visit within 6 months.
5. Clinical decision made to initiate treatment with lifitegrast ophthalmic solution prior to enrollment in the study.
6. Patient agrees to be included after signing an informed consent.

Exclusion criteria

1. Known hypersensitivity to lifitegrast or its components.
2. Dry eye secondary to scarring or destruction of conjunctival goblet cells.
3. Patients with active or history of ocular herpes and or other ocular infection within the last 30 days.
4. Any contra-indication as per the label.
5. Refusal to give signed informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include newly started DED patients on lifitegrast ophthalmic solution: DED diagnosed patients who did not receive lifitegrast ophthalmic solution during the 6 months prior to the index date; that started lifitegrast ophthalmic solution during the active recruitment period. The patient will be the unit of analysis. This is critical in the inclusion/exclusion and study analysis.
  .
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-07-31 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients attaining 30% improvement of eye dryness from Baseline | Baseline, month 3
  Percentage of patients attaining 30% improvement of eye dryness from Baseline at Month 3 (using the Eye Dryness Score -(EDS)). The EDS is rated using a visual analog scale (VAS) measured on a scale of 0 (no discomfort) to 100 (maximal discomfort).

SECONDARY OUTCOMES:
Percentage of patients describing eye dryness using EDS score | Day 0, Day 1, month 3 and month 6
  Eye Dryness Score (EDS) is rated using a Visual Analogue Scale (VAS) measured on a scale of 0 (no discomfort) to 100 (maximal discomfort)
Percentage of patients describing ocular burning/stinging, ocular pain, foreign body sensation, itching, eye discomfort, photophobia | Day 0, Day 1, month 3 and month 6
  Percentage of patients describing ocular burning/stinging, ocular pain, foreign body sensation, itching, eye discomfort, photophobia will be provided
Percentage of patients describing visual symptoms such as reduced vision, blurred vision, and fluctuation relative to DED | Day 0, Day 1, month 3 and month 6
  Percentage of patients describing visual symptoms such as reduced vision, blurred vision, and fluctuation relative to Dry eye disease (DED) will be provided
Dry Eye Questionnaire-5 (DEQ5) 5-item | Day 0, Day 1, month 3 and month 6
  The DEQ-5 consists of five questions that assess the following: frequency of watery eye, discomfort, and dryness (scored on a 0-4 scale) and late day discomfort and dryness intensity (scored on a 0 -5 scale).
Percentage of DED patients with matrix metalloproteinase-9 (MMP-9) levels | Day 0, Day 1, month 3 and month 6
  Percentage of DED patients with matrix metalloproteinase-9 (MMP-9) levels will be provided. Matrix metalloproteinase 9 is an inflammatory biomarker that has been shown to be elevated in the tears of DED patients. MMP-9 testing is a valuable diagnostic tool in identifying the presence of ocular surface inflammation in DED patients. MMP-9 level results are classified as positive or negative
Tear film break up time (TBUT) | Day 0, Day 1, month 3 and month 6
  Tear film break up time (TBUT) is a clinical test used to assess the evaporative dry eye disease. The TBUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film; a TBUT under 10 seconds is considered abnormal
Schirmer tear test (STT) score | Day 0, Day 1, month 3 and month 6
  Schirmer tear test measures maximal tear secretion capacity by assessing the amount of tears produced on filter paper in 5 minutes, with normal tear production defined as over 10 mm
Conjunctival and corneal staining score | Day 0, Day 1, month 3 and month 6
  The conjunctival and corneal staining score defined by the National Eye Institute grading system which divides the corneal and conjunctival surfaces to measure fluorescein uptake. Each of the 5 areas of the cornea are graded 0 to 3, with Grade 0 specifying no staining is present, for a total maximum score of 15
Dry Eye Severity Level (DESL) | Day 0, Day 1, month 3 and month 6
  Based on either the symptoms or signs that point to severity of the patient, the DESL can be classified as mild, moderate or Severe
DED patients: Number of participants by cause/type of DED | Baseline
  Cause/Type of DED:
  * Meibomian gland dysfunction
  * Graft versus host disease
  * Primary Sjögren's syndrome
  * Secondary Sjögren's syndrome
  * Other
DED patients: Number of participants by ocular diseases | Baseline
  Ocular diseases:
  * Amblyopia
  * Cataract
  * Glaucoma
  * Macular degeneration
  * Previous ocular injury
  * Strabismus
  * Other ocular diseases
DED patients: Number of participants with comorbidities at time of treatment initiation with lifitegrast ophthalmic solution | Baseline
  DED patients: Number of participants with comorbidities at time of treatment initiation with lifitegrast ophthalmic solution will be provided
DED patients: Number of participants by other DED treatments received prior to therapy (concomitant use) with lifitegrast ophthalmic solution | Baseline
  Other DED treatments :
  * Antibiotics (eg, topical, oral)
  * Cequa (cyclosporine ophthalmic solution)
  * Cyclosporine
  * OTC artificial tears
  * Nutraceuticals (eg, fish oil)
  * Restasis (cyclosporine ophthalmic emulsion)
  * Topical corticosteroids
  * Topical cyclosporine
  * Topical cyclosporine with oral tetracycline
  * Others
DED patients: Number of participants by DED-related surgical procedures received prior to lifitegrast ophthalmic solution | Baseline
  DED-related surgical procedures received prior to lifitegrast ophthalmic solution:
  * Punctal plugs
  * Thermal pulsation treatment (eg, intense pulsed light (IPL), iLux™, Lipiflow®)
  * Other DED-related surgical procedures
DED patients: Number of participants with non-ocular medications | Baseline
  DED patients: Number of participants with non-ocular medications will be provided
DED patients: Number of participants by use of contact lenses | Baseline
  Use of contact lenses (report type of contact lenses if available):
  * Daily
  * Disposable soft
  * Extended wear
  * Spherical
  * Toric
  * Other
DED patients: Number of participants by history of ocular surgery | Baseline
  History of ocular surgery:
  * Cataract surgery
  * Corneal surgery
  * Eye muscle surgery
  * Glaucoma surgery
  * Laser eye surgery
  * Oculoplastic surgery
  * Other ocular surgery
DED patients: Percentage of patients with DED baseline severity, symptoms and signs prior to the start of the medication | Baseline
  Percentage of patients with DED baseline severity, symptoms and signs prior to the start of the medication will be provided
DED patients: Total screen time | Baseline
  Total screen time (hours per day).
DED patients: Number of patients wearing a mask | Baseline
  Wearing a mask (hours per day).
DED patients: Time to treatment discontinuation | Month 6
  DED patients: Time to treatment discontinuation will be provided. Treatment discontinuation is defined as the time from the index date (date of initiation of lifitegrast ophthalmic solution) until the earliest of treatment discontinuation or end of the study period.
DED patients: Reason for discontinuation | month 6
  DED patients: Reason for discontinuation will be provided if available
DED patients: Time to add-on therapy of lifitegrast ophthalmic solution to Restasis | month 6
  Time to add-on therapy of lifitegrast ophthalmic solution to Restasis (cyclosporine ophthalmic emulsion) and vice versa during the first 6 months of treatment
DED patients: Percentage with treatment switch from lifitegrast ophthalmic solution | month 6
  Percentage of DED patients with treatment switch from lifitegrast ophthalmic solution to other DED solutions (eg, Restasis (cyclosporine), OTC artificial tears, topical corticosteroids, antibiotics, nutraceuticals) during the first 6 months of treatment
DED patients: Percentage of patients with add-on therapy of lifitegrast ophthalmic solution to Restasis | month 6
  Percentage of DED patients with add-on therapy of lifitegrast ophthalmic solution to Restasis (cyclosporine ophthalmic emulsion) and vice versa during the first 6 months of treatment
DED patients: Percentage of patients in treatment with lifitegrast ophthalmic solution plus other DED non-therapeutic solutions | month 6
  Percentage of DED patients in treatment with lifitegrast ophthalmic solution plus other DED non-therapeutic solutions (eg, OTC artificial tears, topical corticosteroids, antibiotics, nutraceuticals) during the first 6 months of treatment
DED patients: Percentage of patients with occurrence of the following DED-related surgical procedures following initiation of lifitegrast ophthalmic solution | month 6
  Percentage of DED patients with occurrence of the following DED-related surgical procedures following initiation of lifitegrast ophthalmic solution during the first 6 months of observation:
  * Punctual plugs
  * Thermal pulsation treatment (IPL, iLux, Lipiflow)
  * Other DED-related surgical procedures (eg, amniotic membrane placement)
Number of DED-related clinic visits (public or private) | 6 months
  Number of DED-related clinic visits (public or private) during the 6 months of observation
Number of days absent from work during the 6 months follow-up | Baseline, month 6
  Number of days absent from work (absenteeism) during the 6 months follow-up. This will be measured using the Work Productivity and Activity Impairment (WPAI) questionnaire at Baseline and at 6 months.
  The Work Productivity and Activity Impairment: Specific Health Problem (WPAI: SHP) is a 6-item questionnaire that assesses work performance and daily activities performance. The WPAI scores productivity by measuring absenteeism (work time missed), presenteeism (impairment at work/reduced on-the-job effectiveness), work productivity loss (overall work impairment/absenteeism plus presenteeism), and impairment of daily activities (i.e., work around the house, shopping, exercising, childcare, studying). WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity,

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No